CLINICAL TRIAL: NCT06940375
Title: Construction of Prediction Models for Metabolic - Associated Fatty Liver Disease and Liver Fibrosis in HIV - Infected Individuals
Brief Title: Incidence of Liver Disease-Related Outcomes in People With HIV
Acronym: PWH
Status: Recruiting | Type: Observational
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Yinzhong Shen, Clinical Professor, Shanghai Public Health Clinical Center
Other Study IDs: GKT1190; SHDC22024317 (Other Grant/Funding Number: Shanghai Hospital Development Center)
Record Dates: First submitted 2025-03-21; First posted 2025-04-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: MAFLD; Liver Fibrosis; MASH; HIV; Hepatic Steatosis; Metabolic Syndrome (MetS)
Keywords: people with HIV; metabolic associated fatty liver disease; liver fibrosis; prognosis
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Ten milliliters of fasting blood samples will be collected for the extraction of whole blood, plasma and peripheral blood mononuclear cells (PBMCs) to meet research requirements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Abdominal ultrasound , Fibroscan and body composition analysis examination — Abdominal ultrasound and Fibroscan examinations were conducted to obtain LSM, CAP, and calculate the FAST score. Bioelectrical impedance analysis was performed to obtain the content of subcutaneous and visceral fat.
  Other Names: TE; BIA

SUMMARY:
Antiretroviral therapy can effectively control the replication of HIV, prolong the lifespan of patients infected with HIV, and improve their quality of life.At the same time, non-AIDS-related diseases such as diabetes and chronic liver diseases are increasing day by day.Metabolic associated fatty liver disease (MAFLD) is a chronic progressive liver disease caused by overnutrition and insulin resistance in genetically susceptible individuals. It was formerly known as non-alcoholic fatty liver disease (NAFLD).With the continuous improvement of living standards and the constant change of lifestyles, the incidence of metabolic associated fatty liver disease is gradually increasing. Metabolic associated steatohepatitis (MASH) may further develop into liver cirrhosis, liver failure and hepatocellular carcinoma, and is the third most common cause of liver transplantation.

In HIV patients, early identification of significant liver fibrosis and MASH with fibrosis is of vital importance.However, due to the fact that the pathogenesis of liver fibrosis in HIV patients is more complex than that in the general population, it involves multiple factors such as the virus, reverse transcriptase drugs, chronic inflammation, and immune disorders.However, the current clinical research on metabolic-related fatty liver fibrosis in people with HIV is still rather limited.

DETAILED DESCRIPTION:
Chronic liver injury caused by various etiologies can lead to liver fibrosis. Liver fibrosis refers to the imbalance between the synthesis and degradation of extracellular matrix in the liver under the influence of various pathogenic factors (viruses, ethanol, autoimmunity, steatosis). For HIV patients, the causes of liver fibrosis are more complex. Firstly, the impact of HIV infection itself, including chronic inflammation and immune activation caused by HIV.Secondly, the liver toxicity side effects of antiretroviral drugs and the immune reconstitution inflammatory syndrome that occurs in some patients at the beginning of treatment, causing liver inflammation and fibrosis.Third, combine various liver diseases-induced fibrosis, including metabolic associated fatty liver fibrosis, etc.In HIV patients, early identification of significant liver fibrosis and MASH with fibrosis is of vital importance. APRI and FIB-4 are currently widely used non-invasive methods for assessing the severity of liver fibrosis.However, due to the more complex pathogenesis of liver fibrosis in HIV patients compared to the general population, the accuracy of APRI and FIB-4 in diagnosis may be affected. Recently, the Fibroscan - aspartate aminotransferase (FAST) score was established to identify high-risk patients with significant liver fibrosis (F2-F4) associated with metabolic associated steatohepatitis (MASH). The FAST score was calculated using the controlled attenuation parameter (CAP), liver stiffness measurement (LSM), and aspartate aminotransferase (AST) level. Moreover, the FAST score has been validated in global clinical trials targeting metabolic associated steatohepatitis.However, in HIV-infected individuals, clinical trials targeting metabolic-associated fatty liver fibrosis are still lacking, and there is a lack of prognostic data for patients with HIV combined with MAFLD.

This is a prospective supplementary follow-up study of HIV patients with MAFLD based on a 5-year retrospective cohort. The investigators aim to explore the incidence of the progression of MAFLD, evaluate the prognostic value of the FASTscore in predicting liver - related and extra - hepatic outcomes among PWH. Additionally, the investigators intend to integrate this with metabolomics to construct prediction models for MAFLD that are suitable for HIV - infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years old
2. HIV positive individuls
3. Had abdominal ultrasound and Fibroscan done between December 2019 and April 2020, with available data of LSM and CAP, and had routine follow - up at our hospital's outpatient department from April 2020 to April 2025.

Exclusion Criteria:

1. Men with excessive alcohol consumption (more than 210g/week) and women with excessive alcohol consumption (more than 140g/week).
2. Suffering from other liver diseases, such as viral hepatitis, drug-induced liver disease, autoimmune liver disease, decompensated liver cirrhosis, liver malignancy, or having had a liver transplantation.
3. Pregnant women and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically diagnosed HIV
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who progress from non - MASH at risk to MASH at risk | Baseline
  Patients will be divided into three groups based on the different severity characteristics of metabolic-associated fatty liver disease (MAFLD). One group consists of patients with non - metabolic - associated fatty liver. Another group is composed of patients with metabolic - associated fatty liver but not at risk of metabolic (dysfunction) - associated steatohepatitis (MASH). The last group is the one at risk of MASH. The diagnosis of metabolic - associated fatty liver disease (MAFLD) is based on abdominal ultrasound, Fibroscan, and metabolic status. A cutoff of FAST>0.35 is used to define MASH at risk.
Number of patients who progress from non - MAFLD to MAFLD | Baseline
  Patients will be divided into three groups based on the different severity characteristics of metabolic-associated fatty liver disease (MAFLD).
  One group consists of patients with non - metabolic - associated fatty liver. Another group is composed of patients with metabolic - associated fatty liver but not at risk of metabolic (dysfunction) - associated steatohepatitis (MASH). The last group is the one at risk of MASH.
  The diagnosis of metabolic - associated fatty liver disease (MAFLD) is based on abdominal ultrasound, Fibroscan, and metabolic status.
  A cutoff of FAST>0.35 is used to define MASH at risk.

SECONDARY OUTCOMES:
Number of participants with cardiovascular events | Baseline
  cardiovascular events include myocardial infarction, arrhythmia and heart failure
Number of participants with extrahepatic tumors | Baseline
  these will be assessed as open-ended questions

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Patient Privacy Issues

REFERENCES:
- [Result] Newsome PN, Sasso M, Deeks JJ, Paredes A, Boursier J, Chan WK, Yilmaz Y, Czernichow S, Zheng MH, Wong VW, Allison M, Tsochatzis E, Anstee QM, Sheridan DA, Eddowes PJ, Guha IN, Cobbold JF, Paradis V, Bedossa P, Miette V, Fournier-Poizat C, Sandrin L, Harrison SA. FibroScan-AST (FAST) score for the non-invasive identification of patients with non-alcoholic steatohepatitis with significant activity and fibrosis: a prospective derivation and global validation study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):362-373. doi: 10.1016/S2468-1253(19)30383-8. Epub 2020 Feb 3. PMID 32027858
- [Result] Cervo A, Shengir M, Patel K, Sebastiani G. NASH in HIV. Curr HIV/AIDS Rep. 2020 Dec;17(6):601-614. doi: 10.1007/s11904-020-00531-0. PMID 32984925
- [Result] Kaspar MB, Sterling RK. Mechanisms of liver disease in patients infected with HIV. BMJ Open Gastroenterol. 2017 Oct 26;4(1):e000166. doi: 10.1136/bmjgast-2017-000166. eCollection 2017. PMID 29119002
- [Result] Rivera CG, Otto AO, Zeuli JD, Temesgen Z. Hepatotoxicity of contemporary antiretroviral drugs. Curr Opin HIV AIDS. 2021 Nov 1;16(6):279-285. doi: 10.1097/COH.0000000000000706. PMID 34545037
- [Result] Fan JG, Xu XY, Yang RX, Nan YM, Wei L, Jia JD, Zhuang H, Shi JP, Li XY, Sun C, Li J, Wong VW, Duan ZP; Chinese Society of Hepatology, Chinese Medical Association. Guideline for the Prevention and Treatment of Metabolic Dysfunction-associated Fatty Liver Disease (Version 2024). J Clin Transl Hepatol. 2024 Nov 28;12(11):955-974. doi: 10.14218/JCTH.2024.00311. Epub 2024 Nov 4. PMID 39544247
- [Result] Navarro J. HIV and liver disease. AIDS Rev. 2022;25(2):87-96. doi: 10.24875/AIDSRev.M22000052. PMID 35901073
- [Result] Acquired Immunodeficiency Syndrome Professional Group, Society of Infectious Diseases, Chinese Medical Association; Chinese Center for Disease Control and Prevention. Chinese guidelines for the diagnosis and treatment of human immunodeficiency virus infection/acquired immunodeficiency syndrome (2024 edition). Chin Med J (Engl). 2024 Nov 20;137(22):2654-2680. doi: 10.1097/CM9.0000000000003383. Epub 2024 Nov 18. PMID 39602327
- [Result] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines on the management of metabolic dysfunction-associated steatotic liver disease (MASLD). J Hepatol. 2024 Sep;81(3):492-542. doi: 10.1016/j.jhep.2024.04.031. Epub 2024 Jun 7. PMID 38851997